CLINICAL TRIAL: NCT06320236
Title: Emergency Medicine Pulmonary Embolism Testing Multicentre Study
Acronym: EMPET
Status: Recruiting | Type: Observational
Sponsor: Dr. Kerstin de Wit (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Kerstin de Wit, Clinician Investigator Program Director & Research Director for the Department of Emergency Medicine, Queen's University, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 4603
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Embolism; D-dimer; Diagnosis
Keywords: D-dimer; Pulmonary Embolism; Adjust-Unlikely; Diagnostic; Emergency Medicine
MeSH Terms: conditions — Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency department patients tested for pulmonary embolism.
  Interventions: Diagnostic Test: Adjust-Unlikely

INTERVENTIONS:
Diagnostic Test: Adjust-Unlikely — Pulmonary embolism will be excluded during emergency department assessment by the combination of:
  1. 'Pulmonary embolism is the most likely diagnosis' as per the treating physician AND a D-dimer result < 500 ug/L fibrinogen equivalent units;
  2. 'Pulmonary embolism is not the most likely diagnosis' AND D-dimer < age-adjusted threshold; or,
  3. A negative computed tomography scan, planar ventilation perfusion scan or ventilation perfusion-SPECT.
  Emergency departments will use their local laboratory D-dimer assay.

SUMMARY:
It is important to diagnose pulmonary embolism in a timely manner to prevent death and long-term disability. More than half a million people (4-5% of emergency department patients) are tested for pulmonary embolism, although the positive rate is low. Imaging for PE testing exposes patients to radiation, is expensive, adds time to the emergency visit, and can lead to a false positive diagnoses. Existing protocols aimed at reducing unnecessary pulmonary embolism imaging are complex and seldom used by emergency physicians. Too many patients undergo unnecessary pulmonary embolism imaging.

A new tool (called Adjust-Unlikely) could safely reduce pulmonary embolism imaging in Canada. A research group composed of researchers, emergency physicians, and patients developed the Adjust-Unlikely clinical decision rule: a rule which has been customized for emergency physicians and emergency patients. Adjust-Unlikely is highly sensitive at the bedside, meaning there are very few false negative results.

The study aim is to prospectively validate Adjust-Unlikely pulmonary embolism testing in emergency patients with suspected pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient who is tested by an emergency physician for PE

Exclusion Criteria:

* Patient is < 18 years of age
* No documentation of whether PE is the most likely diagnosis
* D-dimer is not tested or else not resulted during the emergency visit
* The D-dimer level is known before documentation of whether PE is the most likely diagnosis
* The D-dimer is ordered prior to the physician assessing the patient
* The patient has previously registered that they opt out of all research at the participating site
* The patient leaves against medical advice
* The patient has had PE or deep vein thrombosis imaging (CT pulmonary angiogram, ventilation-perfusion scan or lower limb ultrasound) within prior 30 days
* There is a new (non-PE) indication for anticoagulation
* The patient was initiated on treatment for presumed PE prior to PE testing
* The patient has previously been enrolled into the study
* The patient has a prior history of lower extremity deep vein thrombosis without availability of a baseline ultrasound scan
* The patient was transferred from another hospital organization
* The patient does not reside in Ontario
* The patient has no valid Ontario Health Insurance Plan card

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patient who is tested by an emergency physician for PE.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of venous thrombosis events | 30 days

SECONDARY OUTCOMES:
Number of venous thrombosis | 90 days
Index presentation Adjust-Unlikely testing results | 90 days
  Positive or negative 'Adjust-Unlikely' testing result

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin de Wit, MD, Principal Investigator — Queens University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No